CLINICAL TRIAL: NCT00245986
Title: Pharmacogenetics of Efavirenz Metabolism: Association of CYP2B6 Genotype and Prolonged Drug Exposure
Brief Title: Effect of Genetics on Metabolism of Efavirenz
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060006; 06-CC-0006
Record Dates: First submitted 2005-10-27; First posted 2005-10-28 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-05-20

CONDITIONS: Metabolism
Keywords: Pharmacokinetics; Cytochrome P450; HIV Resistance; Drug Interaction; Non-Nucleoside Reverse Transcriptase Inhibitors; HIV Positive; Healthy Volunteer; HV
MeSH Terms: conditions — HIV Seropositivity | interventions — Blood Specimen Collection

INTERVENTIONS:
Procedure: Blood draw

SUMMARY:
This study will evaluate the effects of genetics on metabolism of the anti-HIV medicine efavirenz (Sustiva) and will see if Efavirenz interacts with bupropion (Zyban or Wellbutrin), a drug commonly used to treat depression and to help people quit smoking. Efavirenz is metabolized by an enzyme called CYP2B6, which is thought to be more active in some people than in others, depending on their genetic makeup. The rate of metabolism of the drug can affect how the body responds it and perhaps the ability of the HIV virus to develop resistance to it.

Healthy volunteers between 18 and 55 years of age who are non-smokers and HIV-infected men and women 18 years of age and older who are taking efavirenz along with two or three nucleoside reverse transcriptase inhibitors may be eligible for this study. Candidates are screened with a medical history and physical examination and blood tests, including tests to determine which genes they have for four different proteins or enzymes (CYP2B6, CYP3A4, CYP3A5, and MDR1) that metabolize drugs.

Participants are assigned to one of three groups for the following procedures:

-HIV-infected individuals: Blood samples are drawn to measure efavirenz levels, as follows: On the last day of taking efavirenz, the subject skips his or her usual evening efavirenz dose the night before sampling. The next morning at clinic, a catheter (flexible plastic tube) is inserted into a vein in the subject's arm for collecting blood samples. After the first sample is drawn, the subject takes a dose of efavirenz. Eight more blood samples are collected at 1, 2, 4, 6, 8, 12, 24 and 48 hours after taking the efavirenz tablet. (The catheter is removed after the 12-hour sample and the subject is discharged home, and then returns to the clinic for the 24- and 48-hour samples, which are collected through a needle inserted into an arm vein.) The subject returns to the clinic four more times for a single blood draw at 7, 14, 21 and 28 days after stopping efavirenz.

HIV-infected patients whose HIV viral load reaches 1,000 copies/L or more within 12 months after completing the study are asked to return to the clinic for a blood draw to check the genotype of the virus for drug resistance.

* Healthy Volunteers - Group 1: Blood samples are drawn to measure efavirenz levels, as follows: Participants take one efavirenz tablet once a day for 13 to 15 days. On the last day of taking efavirenz, the subject takes his/her last dose of efavirenz in clinic, where blood is then collected as described above for HIV-infected individuals.
* Healthy Volunteers - Group 2: A catheter is inserted into a vein in the subject's arm and a blood sample is drawn through the catheter. The subject then takes a single bupropion tablet and additional blood samples are drawn at 1,2, 2.5, 3, 3.5, 4, 6, 8, 12, 24 and 48 hours after the dose to measure the amount of drug in the blood. Subjects begin taking efavirenz 0 to 6 days after the last bupropion blood level is measured. As above, subjects will take one efavirenz tablet once a day for 13 to 15 days. On the last day of taking efavirenz, a catheter is inserted into the subject's arm. Two blood samples are drawn through the catheter, the subject takes the daily dose of efavirenz along with a bupropion tablet. Eleven additional blood samples are drawn at 1, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, and 48 hours after taking the pills to measure blood levels of bupropion. Eight additional samples are collected at 1, 2, 4, 6, 8, 12, 24, and 48 hours to measure efavirenz blood levels. (The catheter is removed after the 12-hour sample and the subject is discharged home; the 24- and 48-hour samples are collected through a needle inserted into an arm vein.)

DETAILED DESCRIPTION:
Efavirenz (EFV) is a non-nucleoside reverse transcriptase inhibitor (NNRTI) with a long half-life, allowing for once-daily dosing. Although it is generally well-tolerated and widely used, a major disadvantage of EFV is its relatively low barrier to resistance. The single K103N mutation confers high-level resistance to EFV, as well as to all other NNRTI's. Acquisition of HIV-1 resistance is likely to result from repeated exposure of the virus to subtherapeutic drug concentrations.

When terminating EFV therapy it is recommended that EFV be stopped 1-2 weeks earlier than concomitant antiretrovirals (ARVs) to account for its long washout period. Alternatively, substituting EFV with a protease inhibitor for 1 to 4 weeks has also been recommended. Both strategies attempt to avoid prolonged EFV exposure following discontinuation of concomitant ARVs, thereby lowering the risk of acquiring new resistance mutations. Though widely utilized, neither method has been validated by pharmacokinetic or clinical studies. Genetic differences in CYP2B6 contribute greatly to observed variability in EFV clearance; hence, genetic differences may contribute to significantly different responses to methods of therapy discontinuation. Multiple polymorphisms in CYP2B6 have been identified. Substitutions at positions 516, 785, and 1459 are the most common variants, and appear to be associated with alterations in CYP2B6 activity.

We propose a 2-part study. Part I is to be conducted in HIV-negative volunteers, and consists of: (1) determination of EFV pharmacokinetic (PK) values (following 13-15 days of EFV 600 mg/day) for comparison between CYP2B6 genotypes (including wild-type and allelic variants at positions 516, 785 and 1459), (2) measurement of single EFV plasma concentrations 7, 14, 21, and 28 days after the drug is stopped to assess for differences in EFV exposure between CYP2B6 genotypes, and (3) comparison of bupropion PK values following administration of a single bupropion dose (a) prior to EFV administration and (b) after 13-15 days of EFV, to evaluate whether EFV modulates CYP2B6 metabolism using bupropion as a probe for CYP2B6 function.

Part II is to be conduced in HIV-positive patients who are planning to discontinue (d/c) their EFV therapy, and includes: (1) determination of EFV PK values prior to d/c of therapy for comparison between different CYP2B6 genotypes, (2) measurement of single EFV plasma concentrations 7, 14, 21 and 28 days post-EFV to assess for differences in exposure across CYP2B6 genotypes, and (3) genotypic evaluation of HIV-1 drug resistance performed in any patient with an HIV RNA = 1,000 copies/mL, prior to and after EFV discontinuation (up to 12 months after stopping EFV), as a preliminary study to evaluate the incidence of EFV resistance mutations based on CYP2B6 genotype.

Data from this study will help to describe the relationship between CYP2B6 genetic polymorphisms and the PK variability of EFV, specifically addressing the effect on prolonged EFV exposure following discontinuation of therapy. In addition, this study will determine whether EFV modulates CYP2B6 activity as assessed by bupropion phenotyping. Lastly, it will attempt to provide preliminary information about whether genetic variability in CYP2B6 is related to the incidence of NNRTI-resistance after stopping or changing EFV therapy.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Healthy Volunteers:

Inclusion Criteria:

1. Males and females between the ages of 18 and 55 years.
2. Healthy by medical history and physical exam
3. Laboratory values within established guidelines for participation in clinical studies: AST less than 1.25 x ULN; SCr less than or equal to ULN; hemoglobin equal to or greater than 11 g/dL (for males and females).

5.) Ability to abstain from eating grapefruit or drinking grapefruit juice during EFV administration and EFV PK sampling periods.

6.) Negative serum pregnancy test for females of child-bearing potential (within 1 day before starting EFV).

7.) Females of child-bearing potential who are able and willing to either practice abstinence or use two non-hormonal forms of birth control (such as condoms, diaphragms, IUDs, etc.) while taking EFV and up to the 28th day after their last EFV dose.

8.) Non-smokers for at least 1 month prior to study participation.

Exclusion Criteria:

1. Concomitant routine therapy with any prescription, over-the-counter, herbal, or holistic medications, including oral contraceptives and hormonal IUDs, for 14 days prior to study participation.

   * Intermittent use of acetaminophen and non-steroidal anti-inflammatory medications (i.e. ibuprofen) will be allowed during the study, but should not be taken on the days of pharmacokinetic blood sampling. Intermittent use of the non-sedating antihistamines fexofenadine and cetirizine and topical hydrocortisone cream will be allowed during the study under the supervision of and with the approval of the study team; however, fexofenadine and cetirizine should not be taken on the days of pharmacokinetic blood sampling.
   * A daily multivitamin with minerals will be allowed during the study.
2. Inability to obtain venous access for blood sample collection.
3. The presence or history of any of the following: HIV infection, active tuberculosis, renal disease (chronic or acute renal failure or insufficiency), diabetes, hepatitis B or C infection (as assessed by patient interview) or hepatic impairment, pancreatitis, peptic ulcer disease requiring maintenance pharmacologic therapy, injection drug use, epilepsy or seizure disorders, history of head trauma, any psychiatric illness or symptoms (including, but not limited to depression, bipolar disorder, a history of suicide attempts or suicidal ideation, psychosis, schizophrenia, and bulimia or anorexia nervosa) as assessed by patient interview and through clinician evaluation using the Beck Depression Index, or any other condition that may interfere with the interpretation of the study results or not be in the best interest of the subject in the opinion of the investigators.
4. Positive pregnancy test or breastfeeding female.
5. A previously documented history of persistent diarrhea or malabsorption that would interfere with the subject's ability to absorb drugs.
6. Drug or alcohol abuse that may impair safety or adherence or interfere with the study results (more than 3 alcoholic drinks per day on a regular basis).
7. History of intolerance or allergic reaction to efavirenz (Sustiva® (Registered Trademark)) or bupropion (Wellbutrin® (Registered Trademark)).

HIV-infected volunteers:

Inclusion Criteria

1. HIV-positive males and females at least 18 years old.
2. On a standard EFV-containing regimen (EFV + 2 or 3 NRTIs) for at least 1 month prior to study participation.
3. Laboratory values within established guidelines for participation in clinical studies53: AST less than or equal to 1.25 x ULN; SCr less than or equal to ULN; hemoglobin equal to or greater than 11 g/dL (for both males and females).
4. Ability to abstain from eating grapefruit or drinking grapefruit juice during the EFV PK sampling period and for 3 days prior.
5. A negative pregnancy test for women of child-bearing potential.

Exclusion Criteria

1.) Concomitant therapy with a PI or any NNRTI other than EFV for 30 days prior to study participation.

2,) Concomitant therapy with any prescription, over-the-counter, herbal, or holistic medications that are known to interact with EFV or modulate CYP2B6 activity for 14 days prior to study participation.

3.) Inability to obtain venous access for blood sample collection.

4.) The presence of any of the following: Any active opportunistic infection (including, but not limited to tuberculosis, Mycobacterium avium complex, cytomegalovirus, Pneumocystis jiroveci, Cryptococcus neoformans, and esophageal candidiasis), renal disease (chronic or acute renal failure or insufficiency), hepatic impairment, pancreatitis, or any other condition that may interfere with the interpretation of the study results or not be in the best interest of the subject in the opinion of the investigators.

5.) A previously documented history of persistent diarrhea or malabsorption that would interfere with the subject's ability to absorb drugs.

6.) Drug or alcohol abuse that may impair safety or adherence or interfere with the study results.

7.) Non-adherence to efavirenz therapy (regularly misses greater than 1 dose/week)

8.) Positive pregnancy test or breastfeeding female.

9.) Severe or potentially life-threatening adverse event/toxicitiy from efavirenz, such that administration of an additional dose of efavirenz would be unsafe and is deemed unwarranted by the study personnel or the patient's primary physician.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 350
Dates: Start 2005-10-18; Study Completion 2008-05-20

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Haas DW, Fessel WJ, Delapenha RA, Kessler H, Seekins D, Kaplan M, Ruiz NM, Ploughman LM, Labriola DF, Manion DJ. Therapy with efavirenz plus indinavir in patients with extensive prior nucleoside reverse-transcriptase inhibitor experience: a randomized, double-blind, placebo-controlled trial. J Infect Dis. 2001 Feb 1;183(3):392-400. doi: 10.1086/318083. Epub 2000 Dec 29. PMID 11133370